CLINICAL TRIAL: NCT04291495
Title: Evaluation of the Effects of Semen Incubation With ANDROSITOL®DGN on Sperm Motility and Mitochondrial Membrane Potential Before and After Oral Supplementation With Antioxidants and Myo-inositol
Brief Title: Evaluation of the Effects of Semen Incubation With ANDROSITOL®DGN on Sperm Motility and Mitochondrial Membrane Potential
Acronym: Androsi-Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Aldo E. Calogero, Professor, University of Catania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANDENDCATANIA_01
Record Dates: First submitted 2019-06-10; First posted 2020-03-02 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Asthenozoospermia; Mitochondrial Damage
Keywords: Male infertility; Sperm parameters; Mitochondrial membrane potential
MeSH Terms: conditions — Asthenozoospermia; Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANDROSITOL®TEST (Experimental): At least 45 patients (13 for each category: low, medium, and high responders, + 15% of hypothetical drop-outs)
  Interventions: Diagnostic Test: ANDROSITOL®TEST

INTERVENTIONS:
Diagnostic Test: ANDROSITOL®TEST — Sperm incubation with ANDROSITOL®DGN and evaluation of sperm motility and mithocondrial membrane potential

SUMMARY:
Mitochondria is the cellular organelle responsible for the production of the energy necessary to fuel sperm motility. It has been demonstrated that mitochondrial efficiency is correlated to the fertilizing capacity of the spermatozoon and to the production of high quality embryos. Mitochondria efficiency is measured in the laboratory setting by evaluating the mitochondrial membrane potential.

Myo-inositol is the most represented stereoisomer of the family of inositols and is the only one physiologically concentrated within the seminal plasma. It is essential for sperm maturation and motility and its deficiency is also associated to a reduced sperm count. Myo-inositol promotes motility and allows recovering a higher number of sperm cells after swim-up, both in normospermic patients and in patients with altered seminal parameters.

Scientific studies have shown that semen samples treated in vitro with ANDROSITOL®DGN, show an improvement in mitochondrial efficiency that results in an increase in spermatozoa progressive motility. Based on the percentage increase in the progressive motility showed by the spermatozoa after incubation with ANDROSITOL®DGN (ANDROSITOL®TEST), it is possible to subdivide the semen samples into three categories: low, medium, and high responders.

The aim of the study is to evaluate whether the in vitro response of spermatozoa to ANDROSITOL®TEST correlates with the in vivo improvement of seminal parameters after oral treatment with antioxidants and myo-inositol.

DETAILED DESCRIPTION:
Mitochondria is the cellular organelle responsible for the production of the energy necessary to fuel sperm motility. It has been demonstrated that mitochondrial efficiency is correlated to the fertilizing capacity of the spermatozoon and to the production of high quality embryos. Mitochondria efficiency is measured in the laboratory setting by evaluating the mitochondrial membrane potential.

Myo-inositol is the most represented stereoisomer of the family of inositols and is the only one physiologically concentrated within the seminal plasma. It is essential for sperm maturation and motility and its deficiency is also associated to a reduced sperm count. Myo-inositol promotes motility and allows recovering a higher number of sperm cells after swim-up, both in normospermic patients and in patients with altered seminal parameters.

Scientific studies have shown that semen samples, both pathological and normal, treated in vitro with ANDROSITOL®DGN - a concentrate solution (66X) containing 133 mg/ml of myo-inositol - show an improvement in mitochondrial efficiency that results in an increase in spermatozoa progressive motility. Based on the percentage increase in the progressive motility showed by the spermatozoa after incubation with ANDROSITOL®DGN (ANDROSITOL®TEST), it is possible to subdivide the semen samples into three categories: low, medium, and high responders. High responders have worst mitochondrial function and lower fertilizing capacity, and could represent the category of patients most benefiting from supplementary oral therapy with antioxidants and myo-inositol.

The aim of our study is to evaluate whether the in vitro response of spermatozoa to ANDROSITOL®TEST correlates with the in vivo improvement of seminal parameters after oral treatment with antioxidants and myo-inositol. To do this, the investigators will enroll at least 13 patients for each category (low, medium, and high responder at ANDROSITOL®TEST) and they will re-evaluate conventional seminal parameters, mitochondrial function, and response to ANDROSITOL®TEST after three months of oral supplementation with ANDROSITOL® (dietary supplement of myo-inositol, vitamin E, L-carnitine, L-arginine, folic acid and selenium). The investigators hypothesize that, following supplementation, high-responder patients will exhibit the best improvement in seminal parameters, in particular in sperm motility. Furthermore, if the mitochondrial function is fully restored, they should respond less to the ANDROSITOL®TEST and could be reclassified as low responders.

ELIGIBILITY:
Inclusion Criteria:

/

Exclusion Criteria:

- Absolute asthenozoospermia

* Leukocytospermia
* Positive semen culture and/or urethral swab
* Human Papilloma Virus (HPV) DNA in semen
* History of cryptorchidism
* 3rd degree varicocele
* Markedly reduced testicular volume
* Decompensated diabetes mellitus and other systemic diseases leading to oxidative stress (e.g. chronic renal failure, liver failure)
* Altered concentrations of the following hormones: luteinizing hormone (LH), follicle stimulating hormone (FSH), total testosterone, prolactin, 17β-estradiol
* Alcohol and drug abuse
* Heavy cigarette smoke (≥10 cigarettes/day)
* Body Mass Index (BMI) >35 kg/m2

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Response to the ANDROSI-TEST | T0 and T1 (three months)
  Number of poor and high responders to ANDROSI-TEST
Sperm parameters | T0 and T1 (three months)
  Percentage of total and progressive sperm motility and percentage of spermatozoa with high or low mitochondrial membrane potential

SECONDARY OUTCOMES:
Other Sperm parameters (1) | T0 and T1 (three months)
  Sperm concentration (mil/ml) and Sperm total count (mil/ejaculate)
Other Sperm parameters (2) | T0 and T1 (three months)
  Percentage of spermatozoa with normal morphology
Effects after therapy (1) | T1 (three months) and T2 (six months - three months after supplementation withdrawal)
  Re-evaluation of number of poor and high responders to ANDROSI-TEST 3 months after the discontinuation of Andrositol intake
Effects after therapy (2) | T1 (three months) and T2 (six months - three months after supplementation withdrawal)
  Re-evaluation of percentage of total and progressive sperm motility and percentage of spermatozoa with high or low mitochondrial membrane potential 3 months after the discontinuation of Andrositol intake
Effects after therapy (3) | T1 (three months) and T2 (six months - three months after supplementation withdrawal)
  Re-evaluation of sperm concentration (mil/ml) and Sperm total count (mil/ejaculate) 3 months after the discontinuation of Andrositol intake
Effects after therapy (4) | T1 (three months) and T2 (six months - three months after supplementation withdrawal)
  Re-evaluation of Percentage of spermatozoa with normal morphology 3 months after the discontinuation of Andrositol intake

CONTACTS AND LOCATIONS:
Overall Officials: Aldo E. Calogero, Professor, Principal Investigator — University of Catania
Locations (1):
- Department of Clinical and Experimental Medicine, University of Catania, Catania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calogero AE, Gullo G, La Vignera S, Condorelli RA, Vaiarelli A. Myoinositol improves sperm parameters and serum reproductive hormones in patients with idiopathic infertility: a prospective double-blind randomized placebo-controlled study. Andrology. 2015 May;3(3):491-5. doi: 10.1111/andr.12025. Epub 2015 Apr 9. PMID 25854593
- [Background] Condorelli RA, La Vignera S, Di Bari F, Unfer V, Calogero AE. Effects of myoinositol on sperm mitochondrial function in-vitro. Eur Rev Med Pharmacol Sci. 2011 Feb;15(2):129-34. PMID 21434479
- [Background] Condorelli RA, La Vignera S, Bellanca S, Vicari E, Calogero AE. Myoinositol: does it improve sperm mitochondrial function and sperm motility? Urology. 2012 Jun;79(6):1290-5. doi: 10.1016/j.urology.2012.03.005. PMID 22656408
- [Background] Gulino FA, Leonardi E, Marilli I, Musmeci G, Vitale SG, Leanza V, Palumbo MA. Effect of treatment with myo-inositol on semen parameters of patients undergoing an IVF cycle: in vivo study. Gynecol Endocrinol. 2016;32(1):65-8. doi: 10.3109/09513590.2015.1080680. Epub 2015 Sep 11. PMID 26361940
- [Background] Agarwal A, Parekh N, Panner Selvam MK, Henkel R, Shah R, Homa ST, Ramasamy R, Ko E, Tremellen K, Esteves S, Majzoub A, Alvarez JG, Gardner DK, Jayasena CN, Ramsay JW, Cho CL, Saleh R, Sakkas D, Hotaling JM, Lundy SD, Vij S, Marmar J, Gosalvez J, Sabanegh E, Park HJ, Zini A, Kavoussi P, Micic S, Smith R, Busetto GM, Bakircioglu ME, Haidl G, Balercia G, Puchalt NG, Ben-Khalifa M, Tadros N, Kirkman-Browne J, Moskovtsev S, Huang X, Borges E, Franken D, Bar-Chama N, Morimoto Y, Tomita K, Srini VS, Ombelet W, Baldi E, Muratori M, Yumura Y, La Vignera S, Kosgi R, Martinez MP, Evenson DP, Zylbersztejn DS, Roque M, Cocuzza M, Vieira M, Ben-Meir A, Orvieto R, Levitas E, Wiser A, Arafa M, Malhotra V, Parekattil SJ, Elbardisi H, Carvalho L, Dada R, Sifer C, Talwar P, Gudeloglu A, Mahmoud AMA, Terras K, Yazbeck C, Nebojsa B, Durairajanayagam D, Mounir A, Kahn LG, Baskaran S, Pai RD, Paoli D, Leisegang K, Moein MR, Malik S, Yaman O, Samanta L, Bayane F, Jindal SK, Kendirci M, Altay B, Perovic D, Harlev A. Male Oxidative Stress Infertility (MOSI): Proposed Terminology and Clinical Practice Guidelines for Management of Idiopathic Male Infertility. World J Mens Health. 2019 Sep;37(3):296-312. doi: 10.5534/wjmh.190055. Epub 2019 May 28. PMID 31081299
- [Background] Paoli D, Gallo M, Rizzo F, Baldi E, Francavilla S, Lenzi A, Lombardo F, Gandini L. Mitochondrial membrane potential profile and its correlation with increasing sperm motility. Fertil Steril. 2011 Jun;95(7):2315-9. doi: 10.1016/j.fertnstert.2011.03.059. Epub 2011 Apr 20. PMID 21507394
- [Background] Rubino P, Palini S, Chigioni S, Carlomagno G, Quagliariello A, De Stefani S, Baglioni A, Bulletti C. Improving fertilization rate in ICSI cycles by adding myoinositol to the semen preparation procedures: a prospective, bicentric, randomized trial on sibling oocytes. J Assist Reprod Genet. 2015 Mar;32(3):387-94. doi: 10.1007/s10815-014-0401-2. Epub 2015 Jan 20. PMID 25601322
- [Background] Marchetti P, Ballot C, Jouy N, Thomas P, Marchetti C. Influence of mitochondrial membrane potential of spermatozoa on in vitro fertilisation outcome. Andrologia. 2012 Apr;44(2):136-41. doi: 10.1111/j.1439-0272.2010.01117.x. Epub 2011 Jun 30. PMID 21714802
- [Background] Robinson R, Fritz IB. Myoinositol biosynthesis by Sertoli cells, and levels of myoinositol biosynthetic enzymes in testis and epididymis. Can J Biochem. 1979 Jun;57(6):962-7. doi: 10.1139/o79-117. PMID 224990
- [Background] Hinton BT, White RW, Setchell BP. Concentrations of myo-inositol in the luminal fluid of the mammalian testis and epididymis. J Reprod Fertil. 1980 Mar;58(2):395-9. doi: 10.1530/jrf.0.0580395. PMID 7431272
- [Background] Colone M, Marelli G, Unfer V, Bozzuto G, Molinari A, Stringaro A. Inositol activity in oligoasthenoteratospermia--an in vitro study. Eur Rev Med Pharmacol Sci. 2010 Oct;14(10):891-6. PMID 21222378